CLINICAL TRIAL: NCT04407026
Title: Two Novel Peptides Associated With Stage 3 Periodontitis: TFF-1 and TFF-3
Brief Title: Oral and Systemic Levels of TFF-1 and TTF-3 in Periodontal Diseases
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Zeynep Pinar KELES YUCEL, Assistant Prof., Giresun University
Other Study IDs: 2017/009
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid, saliva and serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Healthy control group (n=25) consisted of the volunteers having clinically healthy gingiva, PD≤3 mm, BOP<10% and no sign of clinical attachment loss and radiographic alveolar bone destruction.
  Interventions: Biological: biofluids
- Gingivitis: Gingivitis group (n=25) had PD≤3 mm with BOP>50% in the entire mouth, and no clinical attachment loss or alveolar bone loss.
  Interventions: Biological: biofluids
- Stage 3 periodontitis: Stage 3 periodontitis group included the patients exhibiting PD ≥6 mm and interdental CAL ≥5 mm at %30 or more teeth. They had no more than four teeth loss.
  Interventions: Biological: biofluids

INTERVENTIONS:
Biological: biofluids — Gingival crevicular fluid, saliva and serum samples were obtained.

SUMMARY:
Trefoil factor family (TFF) consists of a group of small peptides that have key roles in host immune response and repair of tissue damage. Interleukin (IL)-1β is a regulatory proinflammatory cytokine in periodontal inflammation. This study aimed to investigate the levels of TFF-1, TFF-3 and IL-1β in gingival crevicular fluid (GCF), saliva and serum of patients with gingivitis, stage 3 periodontitis and healthy individuals.

DETAILED DESCRIPTION:
A total of one hundred participants were enrolled for the study. All individuals were assessed clinically and radiographically. Full-mouth clinical periodontal examinations were performed by the measurements of probing depth (PD), clinical attachment level (CAL), gingival index (GI), plaque index (PI) and bleeding on probing (BOP). All these measurements were recorded at six sites around each tooth with a manual periodontal probe. The participants were categorized into three groups: healthy controls (n=25), patients with gingivitis (n=25) and patients with periodontitis (n=50). Gingival crevicular fluid, saliva and serum samples were collected from each participant one day after the clinical periodontal measurements. TFF-1, TFF-3 and IL-1β levels of these biofluids were determined using the enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* No history of smoking
* Individuals between the ages of 25-50 years
* Having at least 20 natural teeth

Exclusion Criteria:

* Any systemic disorders (i.e. diabetes mellitus, cardiovascular diseases, rheumatoid arthritis, immunological disorders, collagen-metabolic diseases, cancer)
* A history of smoking
* Pregnancy or lactation
* A history of surgical/non-surgical periodontal therapy in the past 1 year
* Drug therapy (e.g. anti-inflammatory, antibiotic treatment or any other pharmacological treatment) in the previous 6 months

Ages: 25 Years to 49 Years | Sex: All
Age Groups: Adult
Study Population: Healthy controls included volunteers with clinically healthy periodontium who had BOP < 10% and PD ≤ 3 mm, no sites with attachment loss or radiographic sign of alveolar bone destruction. Gingivitis patients showed PD ≤ 3 mm with BOP > 50% in the entire mouth as well as no clinical attachment loss or alveolar bone loss. Periodontitis patients (Stage 3) had PD ≥ 6 mm, interdental CAL ≥ 5 mm affecting 30% of the teeth or more and showed radiographic bone loss. They showed also no more than 4 teeth loss due to periodontitis.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid, saliva and serum TFF-1 and TFF-3 levels | one day after the clinical periodontal measurements
  Gingival crevicular fluid, saliva and serum TFF-1 and TFF-3 levels of gingivitis and periodontitis patients as well as healthy individuals were analyzed to identify the potential role of these peptides in periodontal diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Pinar Keles Yucel, Principal Investigator — Giresun University
Locations (1):
- Zeynep Pinar Keles Yucel, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No